CLINICAL TRIAL: NCT00857896
Title: An Open-Label, Dose-Escalating Study Of The Pharmacokinetics, Safety And Tolerability Of Fesoterodine In Pediatric Overactive Bladder Patients Aged 8-17 Years.
Brief Title: Study Of Fesoterodine In Pediatric Overactive Bladder Patients Aged 8-17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0221066
Record Dates: First submitted 2009-02-26; First posted 2009-03-09 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Overactive Bladder; Neurogenic Detrusor Overactivity
Keywords: Study of fesoterodine in pediatric overactive bladder patients
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fesoterodine once daily (Experimental)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — 4 mg once daily for Weeks 1-4 and 8 mg once daily for Weeks 5-8

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics, safety, and tolerability of fesoterodine following administration to pediatric patients, aged 8-17 years, with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* A total body weight >25 kg (55 lbs).
* Symptoms of urinary frequency (average ≥8 daily bathroom visits to urinate) and urgency to urinate, with or without urgency incontinence, for at least 6 months prior to enrolment, OR
* Stable neurological disease and urodynamically confirmed detrusor overactivity, who may require intermittent catheterization for management of urinary drainage.

Exclusion Criteria:

* Treatment with an investigational drug within 4 weeks or 5 half-lives, whichever is longer, before first study dose
* Ongoing use of potent CYP3A4 inhibitors or inducers or CYP2D6 inhibitors
* Ongoing use of another drug for treating overactive bladder
* Uncontrolled narrow angle glaucoma, urinary or gastric retention

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Liberty Township, Ohio

REFERENCES:
- [Derived] Sano Y, Shoji S, Shahin M, Sweeney K, Darekar A, Malhotra BK. Population Pharmacokinetic and Pharmacodynamic Modeling of Fesoterodine in Pediatric Patients with Neurogenic Detrusor Overactivity. Eur J Drug Metab Pharmacokinet. 2023 May;48(3):257-269. doi: 10.1007/s13318-023-00818-8. Epub 2023 Mar 9. PMID 36892754
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221066&StudyName=Study%20Of%20Fesoterodine%20In%20Pediatric%20Overactive%20Bladder%20Patients%20Aged%208-17%20Years

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine: Fesoterodine 4 milligram (mg) tablet once daily (QD) from Baseline to Week 4, escalated to 8 mg tablet QD for Weeks 5 to 8.
Period: Baseline to Week 4
Arm/Group | Fesoterodine
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Week 5 to Week 8
Arm/Group | Fesoterodine
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 13.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Absorption Rate Constant (Ka)
Time Frame: Day 28 and Day 56
Population: Pharmacokinetic (PK) concentration population: randomized and treated participants who had at least 1 concentration during the study.
Measure: Mean (95% Confidence Interval); unit: 1/hour (hr)
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
1/hour (hr) | 0.44 [0.15 to 0.58]

2. Primary Outcome: Apparent Volume of Distribution (VC/F)
Description: The volume necessary to account for the total amount of drug in the body if it were present throughout the body at the same concentration found in the blood. Estimated using non linear mixed effect modeling.
Time Frame: Day 28 and Day 56
Population: PK Concentration
Measure: Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
Liters (L) | 1010.00 [566 to 1232]

3. Primary Outcome: Area Under the Plasma Drug Concentration Time Curve (AUC)
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: Day 28 and Day 56
Population: Not analyzed due to the limited amount of data available.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Fesoterodine
Number analyzed (Participants) | 0

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 28 and Day 56
Population: Not analyzed due to the limited amount of data available.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Fesoterodine
Number analyzed (Participants) | 0

5. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Day 28 and Day 56
Population: Not analyzed due to the limited amount of data available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 0

6. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 28 and Day 56
Population: Not analyzed due to the limited amount of data available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 0

7. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated using non linear mixed effect modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 28 and Day 56
Population: PK Concentration
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
L/hr | 86.70 [63.9 to 98.1]

8. Secondary Outcome: Post-void Residual (PVR) Volume
Description: Volume of urine remaining in the bladder immediately after urination.
Time Frame: Baseline, Week 4, and Week 8 post-dose
Population: Safety Population: all participants who were known to have received study medication; Number of participants analyzed (N) = participants not performing clean intermittent bladder catheterization (CIC); n = participants not performing CIC at specified time point.
Measure: Median (Full Range); unit: mL
Arm/Group | Fesoterodine
Number analyzed (Participants) | 12
mL
  Baseline (n=10) | 6.00 [0.00 to 65.00]
  Week 4 (n=12) | 4.00 [0.00 to 90.00]
  Week 8 (n=8) | 25.00 [0.00 to 70.00]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Fesoterodine 4 mg: Fesoterodine 4 mg tablet QD anytime during the study
- Fesoterodine 8 mg: Fesoterodine 8 mg tablet QD anytime during the study
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/20
Other Adverse Events (participants affected / at risk) | 8/21 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg (N=21) | Fesoterodine 8 mg (N=20)
Constipation (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg (N=21) | Fesoterodine 8 mg (N=20)
Hip dysplasia (Congenital, familial and genetic disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 3
Viral infection (Infections and infestations) | 0 | 1
Residual urine volume increased (Investigations) | 0 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.